CLINICAL TRIAL: NCT04337619
Title: Mindfulness and Acceptance Based Behavioral Treatment for Weight Loss
Brief Title: Project Activate: Mindfulness and Acceptance Based Behavioral Treatment for Weight Loss
Acronym: Activate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Meghan Butryn, Professor, Drexel University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01DK119658 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-04-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss; Behavioral treatment; Acceptance-based behavioral weight loss treatment; Acceptance and Commitment Therapy; Multiphase Optimization Strategy
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Standard Behavioral Weight Loss Treatment (Experimental)
  Interventions: Behavioral: Behavioral Treatment
- Behavioral + Mindful Acceptance (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Mindful Acceptance
- Behavioral + Values (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Values
- Behavioral + Mindful Awareness (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Mindful Awareness
- Behavioral + Acceptance + Values (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Mindful Acceptance; Behavioral: Values
- Behavioral + Acceptance + Awareness (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Mindful Acceptance; Behavioral: Mindful Awareness
- Behavioral + Values + Awareness (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Values; Behavioral: Mindful Awareness
- Behavioral + Acceptance + Values + Awareness (Experimental)
  Interventions: Behavioral: Behavioral Treatment; Behavioral: Mindful Acceptance; Behavioral: Values; Behavioral: Mindful Awareness

INTERVENTIONS:
Behavioral: Behavioral Treatment — Standard Behavioral Weight Loss Treatment (remotely delivered)
Behavioral: Mindful Acceptance — Integration of acceptance and willingness skills into Standard Behavioral Weight Loss Treatment (remotely delivered).
  Arms: Behavioral + Acceptance + Awareness; Behavioral + Acceptance + Values; Behavioral + Acceptance + Values + Awareness; Behavioral + Mindful Acceptance
Behavioral: Values — Integration of values clarification and awareness skills into Standard Behavioral Weight Loss Treatment (remotely delivered).
  Arms: Behavioral + Acceptance + Values; Behavioral + Acceptance + Values + Awareness; Behavioral + Values; Behavioral + Values + Awareness
Behavioral: Mindful Awareness — Integration of mindfulness and present-moment awareness skills into Standard Behavioral Weight Loss Treatment (remotely delivered).
  Arms: Behavioral + Acceptance + Awareness; Behavioral + Acceptance + Values + Awareness; Behavioral + Mindful Awareness; Behavioral + Values + Awareness

SUMMARY:
Mindfulness and Acceptance based Behavioral Therapies (MABTs) are among the most promising behavioral approaches for obesity, with two recent large trials showing that they achieve better initial weight loss and/or better weight loss maintenance than does gold standard BT. However, results vary, potentially due to inconsistencies in how MABT components are utilized and emphasized. Optimizing MABTs using a typical approach, i.e., successive randomized controlled trials of various MABT packages, is slow and difficult. Multiphase Optimization Strategy (MOST) has been developed as a better method of optimizing treatment. Consistent with Phase I of MOST, we derived three MABT components from the theoretical literature. Evaluation of MABT components through a factorial design (MOST Phase II) will allow us to determine the independent and interacting efficacies of each MABT component, in addition to the identification of subsets of individuals most or least responsive to each component. Whereas mediational analyses have been inconclusive, the use of a factorial design will allow for a critical test of the main and interaction effects of individual MABT treatment components. The current study will use a full factorial design to identify the independent and combined effects of three core MABT components (Awareness, Acceptance, and Values Clarity) as additions to remotely delivered weight loss counseling. Moderators of treatment outcome (disinhibited eating, food cue susceptibility, emotional eating, delay discounting, and inhibitory control), and mediator/process variables implicated in MABTs (mindful eating, acceptance of food cues, mindfulness, body responsiveness, autonomous motivation, values clarity, hunger/satiety perceptions, and motivation and pleasure resulting from social functioning) will be assessed as well.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be of overweight or obese BMI (27-50 kg/m2)
* Individuals must be adults (aged 18-70)
* Completion of a 3-day food diary
* Completion of baseline assessment tasks
* Willingness to lose weight, be physically active, and participate in-group sessions.
* Participants must also provide consent for the research team to contact their personal physician if necessary to provide clearance or to consult about rapid weight gain.

Exclusion Criteria:

* Inability to engage in physical activity (defined as walking a city block without stopping)
* Medical or psychiatric condition that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to comply with the program
* Recently began or changed the dose of a medication that can cause significant change in weight
* History of bariatric surgery; weight loss of > 5% in the previous 3 months
* Currently pregnant or breastfeeding or planning to become pregnant
* Planning to, or participating in, another weight loss treatment in the next 3 years.
* Engaging in compensatory vomiting, other severe compensatory behaviors, or more than 12 of any compensatory behavior in the previous 3 months
* Experiencing significant loss of control eating (9 or more binge episodes in the previous 3 months)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

PRIMARY OUTCOMES:
Weight change | Measured at baseline, mid-treatment (6 months), post-treatment (12 months), and at 6-, 12-, and 24-month follow-up (i.e., at 0, 6, 12, 18, 24 and 36 months).
  Measured at home using a standardized weighing procedure. Participants will be weighed in lightweight clothes without shoes using a standardized bluetooth scale accurate to 0.1 kg.

SECONDARY OUTCOMES:
Dietary intake | Measured at baseline, mid-treatment (6 months), post-treatment (12 months), and at 6-, 12-, and 24-month follow-up (i.e., at 0, 6, 12, 18, 24 and 36 months).
  Measured with a 25-item Food Frequency Questionnaire developed by the research team for this study.
Physical activity | Measured at baseline, mid-treatment (6 months), post-treatment (12 months), and at 6-, 12-, and 24-month follow-up (i.e., at 0, 6, 12, 18, 24 and 36 months).
  Measured in minutes per week of moderate-to-vigorous physical activity (MVPA) using the FitBit Charge 2, 3, 4, and 5, consumer-grade wrist-worn activity trackers utilized in several other studies.
Change in quality of life | Measured at baseline, mid-treatment (6 months), post-treatment (12 months), and at 6-, 12-, and 24-month follow-up (i.e., at 0, 6, 12, 18, 24 and 36 months).
  Measured using the Quality of Life Inventory (QOLI).

CONTACTS AND LOCATIONS:
Overall Officials: Evan M Forman, PhD, Principal Investigator — Drexel University Center for Weight, Eating and Lifestyle Science
Locations (1):
- Drexel University Center for Weight, Eating and Lifestyle Science, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chabria R, Hagerman CJ, Crane N, Ehmann M, Knudsen FM, Brown KL, Forman E, Butryn ML. Racial disparities in the efficacy of traditional versus acceptance-based behavioral weight loss. Health Psychol. 2025 Jul 24:10.1037/hea0001537. doi: 10.1037/hea0001537. Online ahead of print. PMID 40705619
- [Derived] Crochiere RJ, Butryn ML, Zhang F, Beaulieu K, Maher JP, Huang Z, Cong C, Forman EM. Intraday relations between physical activity and energy intake among behavioral weight loss participants. Health Psychol. 2024 May;43(5):376-387. doi: 10.1037/hea0001358. Epub 2024 Jan 8. PMID 38190202